CLINICAL TRIAL: NCT01131091
Title: A Phase 1, Multicenter, Open Label, Single Dose Study to Evaluate the Effect of Renal Insufficiency on the Pharmacokinetics of SK 0403
Brief Title: A Multicenter, Open Label, Single Dose Study to Evaluate the Effect of Renal Insufficiency on the Pharmacokinetics of SK 0403
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Roger Morgan, MD Chief Medical Officer, Kowa Research Institute, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SK-0403-1.02US
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Other): Subjects with end stage renal disease (ESRD) who are receiving hemodialysis treatment
  Interventions: Drug: SK-0403
- Group B (Other): Subjects with severe renal impairment
  Interventions: Drug: SK-0403
- Group C (Other): Subjects with moderate renal impairment
  Interventions: Drug: SK-0403
- Group D (Other): Subjects with mild renal impairment
  Interventions: Drug: SK-0403
- Group E (Other): Healthy subjects
  Interventions: Drug: SK-0403

INTERVENTIONS:
Drug: SK-0403 — SK-0403 400 mg

SUMMARY:
This is a Phase 1, multicenter, open label, single dose study. A total of 30 subjects are planned (5 groups of 6 subjects each.)

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open label, single dose study. A total of 30 subjects are planned (5 groups of 6 subjects each) as follows:

Group A: Subjects with ESRD who are receiving hemodialysis treatment

Group B: Subjects with severe renal impairment

Group C: Subjects with moderate renal impairment

Group D: Subjects with mild renal impairment

Group E: Healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult male or female aged 18 to 79 years, inclusive.
* All female subjects (that are not 2 years postmenopausal with a documented serum follicle stimulating hormone level >35 mIU/mL) must have a negative serum pregnancy test at Screening and upon Check in to the study clinic.
* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is able and willing to comply with the protocol and study procedures.

Exclusion Criteria:

* Subject has a BMI >37 kg/m2.
* Subject has taken any prescribed systemic or topical medication
* Subject has donated more than 450 mL of blood within 30 days before the start of dosing.
* Subject has received an investigational drug within 30 days before dosing.
* Subject has had any surgery of the gastrointestinal tract likely to affect drug absorption.
* Subject has had a clinically significant illness

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the effect of renal insufficiency on the pharmacokinetics of a single 400 mg dose of SK 0403. | 72 Hours

SECONDARY OUTCOMES:
The secondary objective is to determine the safety and tolerability of a single 400 mg dose of SK 0403 in subjects with renal insufficiency. | 72 Hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando, Florida
  - Minneapolis, Minnesota